CLINICAL TRIAL: NCT04631367
Title: Kukaa Salama (Staying Safe): A Pre-Post Trial of a mHealth Social Group for Increasing COVID-19 Prevention Practices With Urban Refugee and Displaced Youth in Kampala, Uganda
Brief Title: mHealth Intervention for Increasing COVID-19 Prevention Practices With Urban Refugee and Displaced Youth in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: idrc_covid
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Knowledge, Attitudes, Practice; Covid19
Keywords: Uganda; Forcibly displaced youth; mHealth; Water, Sanitation and Hygiene; RANAS (Risks, Attitudes, Norms, Abilities, Self-Regulation); COVID-19
MeSH Terms: conditions — Behavior; COVID-19; Self-Control | interventions — Masks

STUDY DESIGN:
Intervention Model Description: A single arm, pre-test/post-test trial design will be used to evaluate the effectiveness of a RANAS-informed WhatsApp Social Group intervention on uptake of COVID-19 prevention practices (i.e. hand and respiratory hygiene, physical distancing) with displaced/refugee youth in Kampala, Uganda. A control group design is intentionally not used based on recommendations regarding ethical concerns over the potential withholding of any intervention benefits from a vulnerable group (refugee youth living in informal settlements) in the midst of a pandemic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kukaa Salama: mHealth intervention (Experimental): This is a pre-test/post-test trial, therefore all participants will receive the Kukaa Salama mHealth intervention and will be offered a COVID-19 prevention parcel.
  Interventions: Behavioral: Kukaa Salama: mHealth intervention; Device: Face Mask + Soap

INTERVENTIONS:
Behavioral: Kukaa Salama: mHealth intervention — Kukaa Salama is a 8-week social group program of COVID-19 prevention messaging, which includes sending informational SMS once per week and holding secure group discussions on COVID-19 prevention. Weekly SMS messages will focus on COVID-19 knowledge, including information about transmission, hand washing, respiratory hygiene (coughing and sneezing in ways that won't spread germs), face masks, and physical distancing. Participants can also respond to the SMS with any questions about COVID-19, and the study team will respond with further information and/or additional resources. Weekly group chats will be administered using the customized WelTel platform, and will focus on discussions of how participants can apply and practice the information on COVID-19 prevention in their daily lives. Each group chat will be composed of 15-20 participants, and will be facilitated by a research assistant in Kampala as well as a peer navigator.
Device: Face Mask + Soap — Participants will be offered the opportunity to pick up a parcel that contains a face mask, bar of soap, and a small parcel of food from the partner agency YARID.

SUMMARY:
Uganda hosts 1.4 million refugees, making it Sub-Saharan Africa's largest refugee host community and the third largest globally. Adolescents and young people (AYP) comprise half of the world's 70.8 million forcibly displaced persons, yet they are understudied in pandemics, including in COVID-19. Poverty, overcrowded living conditions, and poor sanitation likely elevate forcibly displaced persons' COVID-19 risks by limiting their ability to practice mitigation strategies. There continue to be significant knowledge gaps regarding the implementation and effectiveness of behaviour change interventions on improving COVID-19 prevention practices (i.e. hand and respiratory hygiene, physical distancing). mHealth (healthcare delivered by mobile phones) is cost-effective, aligned with how youth learn and socialize, vital for physical distancing, and has been used for COVID-19 messaging in other low- and middle-income countries. Nested within an ongoing HIV self-testing cluster-randomized trial, this study aims to develop, implement, and evaluate the effectiveness of an mHealth intervention in increasing COVID-19 prevention practices with displaced/refugee AYP aged 16-24 in Kampala, Uganda. Participants will be enrolled in a 8-week mHealth social group intervention program that is informed by the RANAS (Risks, Attitudes, Norms, Abilities, and Self-Regulation) approach to Water, Sanitation, and Hygiene. Using a pre-test/post-test design, this study will assess changes in participants' self-efficacy (e.g. ability, confidence, adherence) in COVID-19 prevention practices.

DETAILED DESCRIPTION:
Background & Objectives: The proposed study will be nested within an ongoing cluster-randomized HIV self-testing trial (Tushirikiane) in Kampala, Uganda. Using a pre-test/post-test design, the proposed study aims to evaluate the effectiveness of a RANAS-informed mHealth intervention on increasing self-efficacy of COVID-19 prevention practices with displaced/refugee youth aged 16-24 in Kampala, Uganda. This research will be conducted in 5 informal settlements ('slums') grouped into 3 clusters based on proximity (1: Kabalanga and Kasanga, 2: Katwe and Nsambya, 3: Rubaga) where most displaced/refugee persons in Kampala live.

Kukaa Salama Intervention: Participants will be invited to take part in a 8-week COVID-19 prevention program; this will involve receiving 1 SMS/week on COVID-19 prevention messaging, delivered using the WelTel secure platform. All SMS will be delivered in participants' language of choice including English, French, Swahili, Luganda, or Kinyarwanda. Participants will also be invited to take part in a weekly group discussion (15 persons/group) using a secure group conversation integration with WelTel. Each week the group discussions will discuss barriers and facilitators and brainstorm solutions to advance COVID-19 prevention. Participants can also ask the research assistant questions by SMS about COVID-19 during Monday-Friday business hours 9 am-5 pm and can also receive psychosocial support from a counselor from Interaid collaborating with the team and YARID. Regardless of participation in the survey or interview, all participants of the parent trial (Tushirikiane) will also be offered a parcel that contains a face mask, a bar of soap, and a small parcel of food from the partner agency YARID.

Participant Recruitment and Retention: Tushirikiane participants will be invited to take part in the COVID-19 supplement of voluntary questions related to COVID-19 (i.e., about knowledge and prevention) and subsequent Kukaa Salama intervention. The participants will be informed the COVID-19 survey and Kukaa Salama intervention is voluntary and will not affect their participation in the larger Tushirikiane study. Community collaborators will facilitate recruitment and retention; peer navigators will use multiple study reminder strategies (e.g. social media, texts) to maintain engagement, and we will utilize existing outreach and services by MARPI, YARID, and community partners.

Research Team Training: This research involves collaborations with the Ministry of Health's Most At Risk Population Initiative (MARPI) clinics and YARID's urban refugee youth empowerment centres in Kampala.

mHealth Training: This research involves a collaboration with WelTel's non-profit agency for the supportive SMS intervention. WelTel will develop an integration to include discussion groups in the SMS communication platform: SMS surveys, COVID-19 updates, and discussion content will be delivered via WelTel's secure platform. WelTel will support consolidated communication capture and streamlined data visualization to support ongoing analysis. Weekly COVID-19 informational SMS will inform the moderated discussion focus. Multiple 'chat' methods are planned, including: 'scenarios' mimicking real-life situations; a 'question box'; sharing COVID-19 mitigation photos; short movies/GIFs (6-8 seconds); 'memes'; songs; and motivational drivers. The peer navigators and research coordinator will review group discussions weekly to publish top responses to incentivize engagement. WelTel staff has already conducted training with the research team and peer navigators as part of the larger trial.

COVID-19 Prevention Practices: Participants will be surveyed at 3 time points (time 1: baseline; time 2: 8 weeks; time 3: 16 weeks). At baseline (time 1), participants will complete a RANAS-informed questionnaire adapted to COVID-19 (i.e., about knowledge and prevention practices). These COVID-19 related questions will be delivered by a research assistant who will enter the survey responses directly into a tablet (survey will be on the Survey CTO secure platform that runs online and offline). Following the 8-week Kukaa Salama intervention, participants will be asked to complete the same survey (time 2) and again at a 4-month follow up (time 3) to examine changes in COVID-19 knowledge, prevention, and impacts after the intervention and over time.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled within the Tushirikiane HIV-self Testing cluster randomized trial
* Live in one of the 5 slum/informal settlement sites (Kabalanga, Kasanga, Katwe, Nsambya Rubaga)
* Identify as a refugee/displaced person or have refugee parents
* Age 16-24 years
* Speak English, Luganda, French, Swahili, or Kinyarwanda
* Own or have access to a mobile phone for the duration of the study

Exclusion Criteria:

* Not currently enrolled in the Tushirikiane HIV-self Testing cluster randomized trial
* Lives outside of 5 selected study sites
* Does not identify as a refugee or does not have refugee parents
* Less than 16 or older than 24 years
* Does not speak English, Luganda, French, Swahili, or Kinyarwanda
* Does not have mobile phone

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in COVID-19 Prevention Practices | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in COVID-19 prevention practices, participants are asked to report on their self-efficacy (i.e. ability, confidence, adherence) to practice hand and respiratory hygiene (i.e. hand washing with soap, face mask usage) and physical distancing.

SECONDARY OUTCOMES:
Changes in COVID-19 Risk Awareness | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in COVID-19 risk awareness, participants are asked to report on their perceived risk and vulnerabilites to COVID-19 as well as as their knowledge of symptoms and severity.
Changes in Attitude towards COVID-19 | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in attitudes towards COVID-19, participants are asked to report on their attitude (i.e. feelings, costs/benefits) towards prevention practices as well as towards COVID-19 testing and potential vaccines.
Changes in COVID-19 Norms | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in COVID-19 norms, participants are asked to report on the percieved behaviours approved by others (i.e. social pressues) towards COVID-19 prevention practices, transmission, and stigma.
Changes in COVID-19 Self-Regulation | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in COVID-19 self-regulation, participants are asked about their action plan for implementing COVID-19 prevention practices.
Changes in Depression | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  Depression outcomes will be assessed using the Patient Health Questionnaire -9 item (PHQ-9). Higher scores mean a worse outcome. Range 0-27.
Sexual and Reproductive Health | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in sexual and reproductive health, participants are asked to report on personal experiences (e.g. intimate partner violence) as well as perceived changes in the community (e.g. violence, access to sexual and reproductive health services).
Food and Water insecurity | Time 1 (1 week), Time 2 (8 week), Time 3 (month 16 week)
  To assess changes in food and water insecurity, participants are asked to report on frequency of insufficient food (i.e. going to bed hungry) and inadequate clean water.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen H Logie, PhD, Principal Investigator — University of Toronto, Canada
Locations (1):
- Factor-Inwentash Faculty of Social Work, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The data collected during this study will not be made publicly available due to the possibility of identifying participants using a combination of common demographic and response characteristics. The data may be made available from the corresponding author on reasonable request and upon completing suitable data sharing agreements.

REFERENCES:
- [Derived] Logie CH, Okumu M, Berry I, McAlpine A, Musoke DK, Hakiza R, Perez-Brumer A, Baral S, Kyambadde P. Multi-method findings on COVID-19 vaccine acceptability among urban refugee adolescents and youth in Kampala, Uganda. Glob Public Health. 2023 Jan;18(1):2185800. doi: 10.1080/17441692.2023.2185800. PMID 36883681
- [Derived] Logie CH, Okumu M, Berry I, Hakiza R, Kibuuka Musoke D, Kyambadde P, Mwima S, Lester RT, Perez-Brumer AG, Baral S, Mbuagbaw L. Kukaa Salama (Staying Safe): study protocol for a pre/post-trial of an interactive mHealth intervention for increasing COVID-19 prevention practices with urban refugee youth in Kampala, Uganda. BMJ Open. 2021 Nov 22;11(11):e055530. doi: 10.1136/bmjopen-2021-055530. PMID 34810193